CLINICAL TRIAL: NCT02389790
Title: A Phase II, Open-label, Multicentre Study to Evaluate the Long-term Safety and Efficacy of MT-1303 in Subjects With Moderate to Severe Active Crohn's Disease Who Have Completed the MT 1303-E13 Study
Brief Title: Extension Study of MT-1303 in Subjects With Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-1303-E14
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — amiselimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MT-1303 (Experimental)
  Interventions: Drug: MT-1303

INTERVENTIONS:
Drug: MT-1303

SUMMARY:
The primary objectives of the study are:

-To evaluate the long-term safety and tolerability of MT-1303 in subjects with moderate to severe active Crohn's Disease（CD）

ELIGIBILITY:
Inclusion Criteria:

* The subject completed 14 week Treatment Period in the double blind MT-1303-E13 study as per Protocol.

Exclusion Criteria:

* Permanent discontinuation of study medication prior to the end of treatment Visit in MT-1303-E13

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events | 36 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- Investigational site, City Name, Czechia
- Investigational site, City Name, France
- Investigational site, City Nmae, Germany
- Investigational site, City Nmae, Hungary
- Investigational site, City Name, Israel
- Investigational site, City Name, Italy
- Investigational site, City Nmae, Japan
- Investigational site, City Name, Netherlands
- Investigational site, City Name, Poland
- Investigational site, City Name, Slovakia
- Investigational site, City Name, Ukraine